CLINICAL TRIAL: NCT00351845
Title: A Clinical Study to Evaluate the Effect of a Modified Carbohydrate Diet on Body Weight in Overweight or Obese Men and Women
Brief Title: Clinical Study to Test the Effects of a Low-Carbohydrate Diet on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Provident Clinical Research (Other)
Responsible Party: Kevin C. Maki, PhD, Provident Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 203470
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Low carbohydrate diet (behavior)

SUMMARY:
The purpose of this study is to test the effects of a modified carbohydrate diet versus a portion controlled diet in overweight or obese men and women on body weight.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age.
* Waist circumference measurement at Visit 1 (week -1) of ³ 87 cm for females and ³ 90 cm for males.
* Subject agrees to discontinue all use of supplements or multivitamins (except for those provided during study period) by Visit 2 (week 0).
* Normally active and judged to be in good health on the basis of medical history and routine laboratory tests.
* Subject must be willing to follow the assigned diet and maintain usual physical activity level throughout the trial.
* Subject understands the procedures and requirements of the study by providing written informed consent and authorization for protected health information disclosure.

Exclusion Criteria:

* Weight loss of > 10 lb in the two months prior to screening.
* Body mass index (BMI) > 37.0 kg/m2.
* Current smoker (any cigarette use) or history of smoking within 6 months prior to screening.
* Postmenopausal women who are current users of hormone therapy or have discontinued hormone therapy within 2 months prior to screening.
* History or presence of significant cardiac, renal, hepatic, pulmonary, biliary, or endocrine disorders.
* Uncontrolled hypertension (systolic blood pressure ³ 160 mm Hg or diastolic blood pressure ³ 100 mm Hg on two consecutive visits).
* History of recurrent nephrolithiasis, or an acute episode of nephrolithiasis within the last year prior to screening.
* History of symptomatic cholelithiasis, unless subject has undergone cholecystectomy.
* History of gastrointestinal surgery for weight-reducing purposes.
* Active gastrointestinal disorders such as peptic ulcer disease or malabsorption syndromes (controlled lactose intolerance or gastroesophageal reflux disease are acceptable.)
* Pancreatic disease: pancreatic enzyme deficiency, history of pancreatitis.
* Fasting blood glucose ≥ 126 mg/dL at visit 1 or diagnosed diabetes mellitus.
* Use of any weight loss medications, supplements, programs, or meal replacement products intended to alter body weight within 4 weeks of the screening visit or during the course of the study. Occasional use of meal replacement bars or shakes as snacks is acceptable.
* History or presence of cancer in the past 2 years, except for successfully resected basal cell carcinoma of the skin.
* Psychiatric disorders requiring medications (i.e., selective serotonin reuptake inhibitors) or which could interfere with the subject's compliance to the requirements of the protocol.
* History or current presence of any diagnosed eating disorders (binge eating, bulimia, history of anorexia).
* Use of systemic corticosteroids, androgens, or phenytoin.
* Use of pseudo-ephedrine during the study period.
* Use of lipid-lowering drugs or supplements, unless dose stable prior to enrollment (2 months prior for drugs, 2 weeks prior for supplements).
* Use of drugs for regulating hemostasis, other than stable dose aspirin.
* Use of thyroid hormones, except stable-dose replacement therapy for ≥ 2 months prior to enrollment.
* Abnormal laboratory test results of clinical significance, including, but not limited to total cholesterol > 300 mg/dL or triglycerides > 400 mg/dL.
* Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are not using an approved method of contraception. A woman is considered to be of childbearing potential unless she is post-hysterectomy, post-tubal ligation, or ³ 1 year postmenopausal.
* Recent history of (within past 12 months) or strong potential for alcohol or substance abuse. Alcohol abuse will be defined as > 14 drinks per week (1 drink = 12 oz beer, 4 oz wine, or 1 ½ oz distilled spirits).
* Participation in another clinical study within 30 days prior to screening visit (week -1).
* Individual has a condition the Investigator believes would interfere with the evaluation of the subject or put the subject at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-04; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Differences between and within modified carbohydrate and portion-controlled (control) diet treatment groups in the change from baseline (week 0) to week 12 and week 36 in body weight. | week 12 and week 36

SECONDARY OUTCOMES:
Differences between and within modified carbohydrate and control diet treatment groups in the change from baseline (week 0) to week 12 and week 36 in body fat mass (FM). | wwek 12 and week 36
Differences between and within modified carbohydrate and control diet treatment groups in the change from baseline (week 0) to week 12 and week 36 in trunk fat. | week 12 and week 36

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Principal Investigator — Radiant Research Chicago